CLINICAL TRIAL: NCT05915260
Title: Cardiac Magnetic Resonance Imaging in Type 2 Diabetes Mellitus: The Næstved/Slagelse/Ringsted Cohort
Brief Title: CMR in T2DM: The NSR Cohort
Status: Enrolling by invitation | Type: Observational
Sponsor: Slagelse Hospital (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-992
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies; Cardiovascular Magnetic Resonance Imaging; Coronary Microvascular Dysfunction; Myocardium; Fibrosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies; Fibrosis | interventions — Echocardiography; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes: This group will be split up into different groups. DM2 with vs. without complications to diabetes DM2 with vs. without albuminuria/nephropathy or autonomic neuropathy or retinopathy or peripheral neuropathy or macrovascular angiopathy
  Interventions: Diagnostic Test: All subjects will undergo cardiac magnetic resonance imaging with gadolinium contrast and with adenosine myocardial perfusion
- sex and age matched control subjects
  Interventions: Diagnostic Test: All subjects will undergo cardiac magnetic resonance imaging with gadolinium contrast and with adenosine myocardial perfusion

INTERVENTIONS:
Diagnostic Test: All subjects will undergo cardiac magnetic resonance imaging with gadolinium contrast and with adenosine myocardial perfusion — This is a observational follow up study accordingly all subjects will undergo the same examinations
  Other Names: Echocardiography; medical interview; general medical examination, BP, HR e.g.; Examination for non cardiac complications to diabetes

SUMMARY:
This study aims to investigate the myocardial phenotype of patients with type 2 diabetes. From 2016-2019 the investigators recruited a cohort of 296 subjects with type 2 diabetes. All subjects underwent clinical examinations including a gadolinium contrast cardiac MRI.

The current study is a clinical follow-up study of the subjects, thus, the investigators will invite all participants to a reevaluation with cardiac MRI.

Additionally, the investigators will aim at recruiting additionally 400 patients with type 2 diabetes.

The aim it to characterize the phenotype of diabetic cardiomyopathy. Uniquely using cardiac MRI we can measure myocardial microvascular function, myocardial localised and diffuse fibrosis in addition to the quantification of myocardial structure and systolic and diastolic function.

ELIGIBILITY:
Inclusion Criteria:

Few and simple, allowing for a broad cohort.

* Male or female fully capable of providing informed consent
* Informed consent
* Age 18-80 (both included)
* T2DM diagnosed at least 3 months prior to inclusion in the study

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Unable to give informed consent
  * Absolute contraindications to CMR
  * Severe claustrophobia
  * Type 1 diabetes mellitus
  * More than trivial paroxysmal atrial fibrillation, i.e. persistent or permanent atrial fibrillation
  * Women of childbearing potential not on acceptable contraception
  * Contraindications to adenosine, e.g. 2nd or 3rd degree AV-block, severe hypotension, long QT-syndrome, unstable angina pectoris, sinus node dysfunction, decompensated heart failure
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Association of myocardial microvascular function in patients with type 2 diabetes with MACE after 5 years | 5 years follow-up
  Myocardial microvascular function is measured by the myocardial perfusion ratio, quantified by cardiac MRI. MACE defined as CVD events (AMI, HF, stable angina, atrial fibrillation, ventricular arytmia), stroke, death
Clinical factors associated with worsening of diabetic cardiomyopathy after 5 years | 5 years follow-up
  Clinical factors :Albuminuria, autonomic neuropathy, retinopathy, HbA1c, hs-CRP.
  Signs of worsening af diabetic cardiomyopathy: Increased myocardial extracellular volume, decreased myocardial blood flow and myocardial perfusion reserve, decreased strain (GLS; GCS, GRS), increasing E/e´, increasing concentri remodeling index(LV mass / LV end-diastolic volume)
Impact of myocardial perfusion and cardiac cardiac output on perfusion in other organs (kidney, spleen, liver) assed by gadolinium contrast magnetic resonance imaging | Baseline and at 5 years follow-up
  Myocardial perfusion measured by myocardial blood flow and myocardial perfusion ratio quantified by cardiac MRI.
The association of pericardial- and epicardial fat with myocardial function and MACE after 5 year | Baseline and at 5 years follow-up
  Myocardial function: LVEF, LV strain (GLS, GCS, GRS), E/e´, myocardial extracellular volume, myocardial perfusion ratio.
  MACE defined as CVD events (AMI, HF, stable angina, atrial fibrillation, ventricular arytmia), stroke, death

SECONDARY OUTCOMES:
Characterization of the progression of diabetic cardiomyopathy over 5 years, including LV+RV function, the coronary microvascular function, the coronary macrovascular function, fibrosis, aortic stiffness, per and epicardial fat, perfusion of other organs | 5 years follow-up
  Using multivariable regression including age, sex, smoking, Hypertension, HbA1c, CRP, blood pressure, albuminuria, autonomic neuropathy, retinopathy factors associated with either progression or regression of diabetic cardiomyopathy will be tested. Progression of diabetic cardiomyopathy will be defined as increasing myocardial extracellular volume, decreasing myocardial perfusion reserve, decreasing strain (GLS, GCS, GRS), increasing E/e´compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Slagelse Hospital, department of cardiology and endocrinology, medicine 2, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: Yes
On request and with the proper approvals
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code